CLINICAL TRIAL: NCT02745002
Title: Assessment of a Novel, Fast and Automatic CT-to-patient Registration Method During Navigated Bronchoscopy and Endobronchial Ultrasound Bronchoscopy (EBUS)
Brief Title: Navigated EBUS and Functional Imaging in Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); SINTEF Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015/1913
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Bronchial Neoplasms
Keywords: Bronchoscopy; Bronchoscopes
MeSH Terms: conditions — Bronchial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- navigated bronchoscopy (Experimental)
  Interventions: Device: navigated bronchoscopy

INTERVENTIONS:
Device: navigated bronchoscopy
  Other Names: position tracked bronchoscope; navigated endobronchial ultrasound (EBUS)

SUMMARY:
Electromagnetic navigation systems have proved feasible for precise intraoperative guiding during videobronchoscopy and endobronchial ultrasound transbronchial needle aspiration (EBUS-TBNA), based on maps made of preoperative CT images. PET--CT, PET--MRI and fMRI can point out malignant lesions.

When fused into a research navigation system, functional imaging can add information of optimal sampling points in lung cancer staging. Correct image registration is then fundamental. This study is a build--on to NCT02493023, assessing the position and image registration accuracy and clinical feasibility of a multimodal image guiding system in patients referred for lung cancer staging by EBUS--TBNA.

DETAILED DESCRIPTION:
A research navigation platform displays the intraoperative position of the endoscope inside the airways, and shows its position in 3D maps made from the patients' own preoperative images (PET-- CT, PET--MRI or fMRI). Images are acquired ahead of study inclusion. The navigation system acquires position data, first from a videobronchoscope, then from an EBUS--scope (same sort of output data acquired from both endoscopes) equipped with a position sensor for electromagnetic tracking.

From intraoperative position data, the accuracy of the image--to--patient registration (for CT, PET--CT, PET--MRI and fMRI) and the navigation system accuracy are calculated.

Electromagnetic navigation fused with available image modalities can be used to navigate directly and precisely to the area with highest suspicion of malignancy. Multimodal image guiding systems with functional imaging may thereby lead to improvements in endoscopic lung cancer staging, f. i. in diagnostic yield, procedure time and safety.

ELIGIBILITY:
Inclusion Criteria:

* referred to thoracic department St Olavs Hospital due to suspicion of lung cancer
* informed consent

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Endoscope position (measured in millimetres from origo in the x, y and z-plane) in 3 dimensional maps from preoperative CT, PET-CT, PET-MRI or fMRI images | 48 hours
  intraoperative positional data of bronchoscope or endobronchial ultrasound scope (EBUS) measured and stored in navigation system software, used for registration and navigation system accuracy calculations

SECONDARY OUTCOMES:
duration of procedure | 48 hours
  time from first entry of endoscope through vocal cords to final withdrawal of endoscope
patient reported satisfaction | 2 hours
  enquiry on patients´ own experience 2 hours after end of navigated bronchoscopy/EBUS procedure
adverse events | 48 hours
  procedure related adverse events or unexpected incidents registrated
Operator reported satisfaction | 48 hours
  Enquiry on main operator´s experience immediately after end of navigated bronchoscopy/EBUS procedure
Diagnostic yield | 48 hours
  Diagnostic success per TBNA sample defined as >40 lymphocytes/high power field as reported by rapid onsite cytologist

CONTACTS AND LOCATIONS:
Overall Officials: Toril A Nagelhus Hernes, prof, Study Director — Department of Circulation and Imaging
Locations (1):
- Department of Thoracic Medicine, St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sorger H, Hofstad EF, Amundsen T, Lango T, Leira HO. A novel platform for electromagnetic navigated ultrasound bronchoscopy (EBUS). Int J Comput Assist Radiol Surg. 2016 Aug;11(8):1431-43. doi: 10.1007/s11548-015-1326-7. Epub 2015 Nov 28. PMID 26615428